CLINICAL TRIAL: NCT00864994
Title: COPD: Transition of Systemic Inflammation Into Multiorgan Pathology (Study 3). (De Effecten Van Ontsteking op Skeletspieren Bij COPD)
Brief Title: Multiorgan Pathology in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Top Institute Pharma (Other)
Collaborators: University Medical Center Groningen (Other); Maastricht University Medical Center (Other); UMC Utrecht (Other); Danone Institute International (Other); GlaxoSmithKline (Industry); Nycomed (Industry); AstraZeneca (Industry)
Responsible Party: Schols, Prof. dr. ir. AMWJ., Maastricht University Medical Center, Dept. of Respiratory Medicine
Other Study IDs: 23475
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Inflammation; Smoking; Multiorgan pathology; Extra pulmonary manifestations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be retained to investigate differences in candidate genes (SNPs) for COPD and CVD between the different groups.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: • 30 healthy subjects with 20 pack years smoking who have no signs of COPD (age 40-75 years)
- 2: • 30 COPD patients with GOLD stage II (age 40-75 years)

SUMMARY:
There is increasing evidence in the literature that COPD should not be considered as a localised pulmonary disorder but as a systemic disease involving pathology in several extra pulmonary tissues. Well characterized systemic features are a chronic low grade systemic inflammation, altered body composition and a skeletal muscle fibre type shift. There are indications that an absolute or relative increase of fat mass puts COPD patients at increased risk for cardiovascular pathology while muscle atrophy is associated with a high prevalence of osteoporosis and with impaired physical function. The origin of systemic inflammation is poorly understood. Both endogenous and exogenous risk factors contribute to systemic inflammation and extra-pulmonary manifestations of COPD.

Overall objective of study 3:

To compare the pattern and severity of the systemic inflammatory profile in relation to skeletal muscle weakness and cardiovascular risk profile in COPD patients with mild to moderate disease compared to non-susceptible smokers.

Specific objectives:

1. To study the relative contribution of pulmonary and extra pulmonary factors on exercise capacity, skeletal muscle function and health status
2. To relate diet, physical activity and cardiovascular risk factors to body composition, skeletal muscle function and exercise capacity status
3. To study the influence of the emphysema phenotype on extra pulmonary pathology in COPD
4. To study muscle fibre type size and composition and to relate muscle oxidative phenotype with insulin sensitivity, inflammation (local and systemic) and molecular signatures of oxidative energy and protein metabolism.

Study design:

Cross-sectional study. Healthy smoking subjects and COPD patients will undergo extensive clinical, metabolic and inflammatory assessment at the university clinics in Groningen, Maastricht and CIRO Horn.

Study population:

Totally 60 subjects will be included

* 30 healthy subjects who after 20 pack years smoking have no signs of COPD (age 40-75 years)
* 30 COPD patients with GOLD stage II (age 40-75 years)

DETAILED DESCRIPTION:
Primary study parameters/outcome of the study:

1. Smoking history and behaviour, diet and physical activity level assessed by questionnaire
2. Extensive lung function and CT scanning of the lung, ECG
3. Candidate genes for muscle dysfunction and CVD risk
4. Body composition (BIA, waist-hip ratio, DEXA-scan)
5. Systemic inflammation
6. Advanced Glycosylated Endproduct (AGE)
7. Glucose tolerance test
8. Risk factors of metabolic syndrome
9. 6 minute walking distance
10. Handgrip strength
11. Skeletal muscle function by isokinetic dynamometry
12. Physical activity level and pattern by accelerometry
13. Muscle oxidative phenotype, fibre cross-sectional area and molecular signatures obtained in vastus lateralis muscle biopsies before and after incremental cycle ergometry

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

* Totally 22 hours will be spend in the hospital during 3 visits
* CT-scanning of the lung is associated with a radiation burden of 0.8-1.6 mSv (dependent of body weight)
* 50 ml peripheral blood (v. cubiti)
* Muscle biopsy may be associated with temporary pain and haematoma
* Drawing of arterial blood from the radial artery rarely leads to bleeding and transitory nerve damage (numb feeling in wrist/hand area).

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75 years
* Age, pack years, FEV1/FVC and FEV1% predicted must fit in one of 2 groups of table 4.3
* Physically and mentally able to undergo the total study protocol
* Written informed consent

Exclusion Criteria:

* Participation in another study
* Alpha-1-antitrypsin deficiency
* Selected grade 1-3 co-morbidity listed in the ACE-27
* Active pulmonary infection like tuberculosis, pneumonia, flue, tracheobronchitis
* Active extra-pulmonary infection like hepatitis A-C, cystitis, gastroenteritis etc.
* Pulmonary diseases like sarcoidosis, IPF, silicosis, hypersensitivity pneumonitis, asthma
* Life threatening diseases like carcinoma, AIDS (including HIV+), acute leukemia etc.
* Medication that may affect the results of the study: NSAID's, immunosuppressive agents like prednisolon, methotrexate, azathioprine, sintrom tablets, askal
* Antibiotic or prednisolon use in the past 2 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Totally 60 subjects will be included
  * 30 healthy subjects with 20 pack years smoking who have no signs of COPD (age 40-75 years)
  * 30 COPD patients with GOLD stage II (age 40-75 years)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Smoking history and behaviour, diet and physical activity level assessed by questionnaire
Extensive lung function and CT scanning of the lung, ECG
Candidate genes for muscle dysfunction and CVD risk
Body composition
Systemic inflammation
Advanced Glycosylated Endproduct (AGE)
Glucose Tolerance Test
Risk factors of metabolic syndrome
6 minutes walking distance
Handgrip strength
Skeletal muscle function by isokinetic dynamometry
Physical activity level and pattern by accelerometry
Muscle oxidative phenotype, fibre cross-sectional area and molecular signatures obtained in vastus lateralis muscle biopsies before and after incremental cycle ergometry

CONTACTS AND LOCATIONS:
Overall Officials: Emiel Wouters, Prof. dr. MD, Principal Investigator — Maastricht University Medical Center, Dept. of Respiratory Medicine
Locations (1):
- Maastricht University Medical Center, Dept. of Respiratory Medicine, Maastricht, Limburg, Netherlands